CLINICAL TRIAL: NCT01715701
Title: Efficacy of Multilevel Thoracic Paravertebral Nerve Blockade to Reduce Postoperative Pain Following Video-assisted Thoracic Surgery
Brief Title: Efficacy of Paravertebral Nerve Blockade to Reduce Pain Following Thoracoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SG2012-003
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paravertebral nerve blockade (Experimental): A multilevel thoracic paravertebral nerve block will be performed by the anaesthesiologist prior to the induction of general anesthesia. Prior to the block, the anaesthesiologist will locate and mark each level and then, infiltrate the skin with lidocaine 2% (0.5-1 mL). Subsequently, using a Tuohy needle 22G, 5 mL of ropivacaine 0.5% will be injected at each level between T4 and T8. At the end of surgery, before skin closure, a multilevel intercostal nerve block will be performed by the surgeon using 5 mL of saline at each level between T4-T8. A PCA device will be installed upon arrival in the recovery room.
  Interventions: Procedure: Paravertebral nerve blockade
- Intercostal nerve blockade (Active Comparator): Prior to the induction of general anaesthesia, a paravertebral block will be simulated by measuring, marking the patient's skin and applying mild pressure at each level (T4-T8). To preserve the blind, the anaesthesiologist will also infiltrate the skin with lidocaine 2% (0.5-1 mL). A multilevel intercostal nerve block will be performed by the surgeon at the end of surgery before skin closure. Five mL of ropivacaine 0.5% will be injected at each level between T4 and T8. A PCA device will be installed upon arrival in the recovery room.
  Interventions: Procedure: Intercostal nerve blockade
- Patient Controlled Analgesia (PCA) (Active Comparator): Prior to the induction of general anaesthesia, a paravertebral block will be simulated by measuring, marking the patient's skin and applying mild pressure at each level (T4-T8). To preserve the blind, the anaesthesiologist will infiltrate the skin with lidocaine 2% (0.5-1 mL). At the end of surgery, before skin closure, a multilevel intercostal nerve block will be performed by the surgeon using 5 mL of saline at each level between T4-T8. A PCA device will be installed upon arrival in the recovery room.
  Interventions: Procedure: Patient Controlled Analgesia

INTERVENTIONS:
Procedure: Paravertebral nerve blockade — Paravertebral nerve blockade using ropivacaine, intercostal nerve blockade using saline and PCA using hydromorphone or morphine.
  Arms: Paravertebral nerve blockade
Procedure: Intercostal nerve blockade — Intercostal nerve blockade using ropivacaine, simulated paravertebral nerve blockade and PCA using hydromorphone or morphine.
  Arms: Intercostal nerve blockade
Procedure: Patient Controlled Analgesia — Simulated paravertebral nerve blockade, intercostal nerve blockade using saline and PCA using hydromorphone or morphine.
  Arms: Patient Controlled Analgesia (PCA)

SUMMARY:
This study is designed to assess:

* The impact of preoperative multilevel thoracic paravertebral nerve blockade compared to intercostal nerve blockade performed at the end of surgery on the intensity of postoperative pain in subjects having a Patient Controlled Analgesia (PCA) device as their primary analgesic modality.
* The incidence of chronic pain at 6 months following video-assisted thoracic surgery.
* The impact of preoperative multilevel paravertebral nerve blockade on patients' quality of life at 6 months following surgery compared to intercostal nerve blockade and to a control group using PCA alone.

Hypothesis:

1. The basic hypothesis of this study is that preoperative thoracic multilevel paravertebral nerve blockade and multilevel intercostal nerve blockade performed at the end of surgery will provide superior postoperative analgesia and lower opioid consumption compared to PCA alone during the first 24 hours following surgery.
2. Preoperative thoracic multilevel paravertebral nerve blockade will reduce the incidence of chronic pain at 6 months following surgery.
3. Preoperative thoracic multilevel paravertebral nerve blockade and multilevel intercostal nerve blockade performed at the end of surgery will shorten the length of stay in the intermediate intensive care unit and shorten the hospital stay.
4. Preoperative thoracic multilevel paravertebral nerve blockade and multilevel intercostal nerve blockade performed at the end of surgery will reduce postoperative pulmonary complications.

DETAILED DESCRIPTION:
Video-assisted thoracoscopy is increasing in popularity. Although it is considered a less invasive treatment than thoracotomy, patients have reported moderate to severe pain of variable duration. Benefits of adequate analgesia no longer need to be demonstrated. Optimal analgesia leads to faster recovery, reduces the risk of postoperative complications, enhances patient's satisfaction and quality of life following surgery. Furthermore, adequate postoperative analgesia may reduce the occurrence of chronic pain. The incidence of chronic pain following thoracoscopic procedures ranges from 20-47%.

The ideal postoperative analgesia regimen for the pain related to thoracoscopy has not been elucidated.

Systemic opioids given through patient-controlled devices (PCA) may be used after thoracoscopic procedures but the analgesic effect can be limited and undesirable side-effects may occur.

Thoracic epidural has emerged as the preferred pain control technique following thoracotomy. However, the role of epidural analgesia after thoracoscopy remains debatable. Side-effects may outweigh the benefits of the technique in the context of minimally invasive surgeries.

Paravertebral blockade is an alternative to epidural analgesia. The duration of pain relief associated with this technique may vary from 4 to 48 hours. Its effectiveness has been shown to be equal or superior to that of epidural analgesia for post-thoracotomy pain. Its popularity for pain management following thoracotomy has promoted its use after thoracoscopic procedures. Preoperative paravertebral blockade could also result in a reduction of chronic pain following surgery.

Intercostal nerve blockade is widely used to alleviate pain following thoracoscopy. This technique is known to provide adequate short-term pain relief.

Both paravertebral and intercostal blocks could be interesting adjuncts to patient-controlled devices for pain management following thoracoscopic procedures.

This study will compare the efficacy of preoperative paravertebral nerve blockade to intercostal nerve blockade performed before skin closure to PCA alone to reduce the intensity of pain following thoracoscopic procedures. All patients will have a PCA device as their primary analgesic modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an elective or emergency thoracoscopic surgery
* Physical status 1-4

Exclusion Criteria:

* Contraindication to paravertebral nerve blockade (coagulopathy, sepsis or local infection at the site of injection, spinal deformity)
* Severe renal or hepatic insufficiency
* A known allergy to local anesthetics, morphine or hydromorphone
* The inability to understand a verbal numerical pain scale (VNPS) despite previous instruction
* Preexisting pain at the site of the surgical incision
* Current use of opioids, anticonvulsants or tricyclic antidepressants
* A recent history of drug or opioid abuse
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Intensity of postoperative pain | From arrival in the recovery room until 48 hours following surgery
  Intensity of postoperative pain using a Verbal Numeric Pain Scale (VNPS) upon the patient's arrival in and discharge from the recovery room and daily thereafter, for a total duration of two postoperative days.

SECONDARY OUTCOMES:
Opioid consumption | From surgery until 48 hours following surgery
Patient's satisfaction with pain relief | From surgery until 48 hours following surgery
  Patient's satisfaction with pain relief will be assessed using a scale from 1 to 4 (1=very dissatisfied, 4=very satisfied)
Incidence of chronic pain | Six months after surgery
  Incidence of chronic pain will be assessed using the Brief Pain Inventory questionnaire (BPI)
Length of stay in the recovery room | From arrival to discharge from the recovery room (an expected average of one hour)
Length of stay in the intermediate intensive care unit | From arrival to discharge from the intermediate intensive care unit (an expected average of one day)
Length of stay in the hospital | From surgery to discharge from the hospital (an expected average of 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Garneau, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada